CLINICAL TRIAL: NCT02835560
Title: Efficacy and Safety of Ilaprazole Based Bismuth-containing Quadruple Regimen for the First-line Treatment of Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Livzon-IY-81149R
Record Dates: First submitted 2016-07-09; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2012-06

CONDITIONS: Helicobacter Pylori Eradication Antibiotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Ilaprazole-based quadruple therapy for 14 days: Ilaprazole 5mg bid
  Interventions: Drug: Ilaprazole antisecretory drug of each quadruple therapy the Ilaprazole -based quadruple therapy
- Active Comparator (Active Comparator): Esoprazole
  Esoprazole-based quadruple therapy for 14 days: Esoprazole 20mg bid
  Interventions: Drug: Esoprazole antisecretory drug of each quadruple therapy Esoprazole-based quadruple therapy

INTERVENTIONS:
Drug: Ilaprazole antisecretory drug of each quadruple therapy the Ilaprazole -based quadruple therapy — Ilaprazole -based quadruple therapy for 14 days: Ilaprazole 5mg bid, Bismuth Potassium Citrate 220mg bid, amoxicillin 1000mg bid, clarithromycin 500mg bid
  Arms: Experimental
Drug: Esoprazole antisecretory drug of each quadruple therapy Esoprazole-based quadruple therapy — Esoprazole -based quadruple therapy for 14 days: Esoprazole 20mg bid, Bismuth Potassium Citrate 220mg bid, Amoxicillin 1000mg bid, Clarithromycin 500mg bid
  Arms: Active Comparator

SUMMARY:
This study compared efficacy and safety of Ilaprazole based bismuth-containing quadruple regimen therapy including Ilaprazole 5mg, Bismuth Potassium Citrate 220mg, Clarithromycin 500mg and Amoxicillin Cap (Amoxicillin) 1000mg BID on the first line eradication treatment of H.pylori.

Participants are defined as persons who have endoscopically confirmed on gastric or duodenal ulcer(including scar stage), gastritis and dyspepsia confirmed to be H.pylori positive patients in the biopsy and UBT test. For 14 days, participants treated as Esoprazole based bismuth-containing quadruple regimen therapy therapy including Esoprazole 20mg, Bismuth Potassium Citrate 220mg, Clarithromycin 500mg and Amoxicillin Cap (Amoxicillin) 1000mg BID. After treatment, the healing rate was evaluated in the UBT test and Biopsy at 49±5days from the first day dosing.

DETAILED DESCRIPTION:
This study compared efficacy and safety of Ilaprazole based bismuth-containing quadruple regimen therapy including Ilaprazole 5mg, Bismuth Potassium Citrate 220mg，Clarithromycin 500mg and Amoxicillin Cap(Amoxicillin) 1000mg BID on the first line eradication treatment of H.pylori.

Participants are defined as persons who have endoscopically confirmed on gastric or duodenal ulcer(including scar stage), gastritis and dyspepsia confirmed to be H.pylori positive patients in the biopsy and UBT test. For 14 days, Participants treated as Esoprazole based bismuth-containing quadruple regimen therapy therapy including Esoprazole 20mg, Bismuth Potassium Citrate 220mg，Clarithromycin 500mg and Amoxicillin Cap (Amoxicillin) 1000mg BID. After treatment, The healing rate was evaluated in the UBT test and Biopsy at 49±5days from the first day dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have endoscopically confirmed on gastric, duodenal ulcer(including scar) or gastritis confirmed to be H.pylori positive patients in the biopsy and UBT test.
* Subject who fully understands conditions of clinical trial.
* Subject who agrees to participate and spontaneously sign the ICF.

Exclusion Criteria:

* Known hypersensitivity to any component of ilaprazole, Amoxicillin and Levofloxacin.
* Subjects who are taking contraindicated medications for experimental and concomitant drug.
* Patients with abnormal levels in the laboratory tests.
* Total Bilirubin, Creatinine> 1.5 times upper limit of normal.
* AST, ALT, Alkaline phosphatase, BUN> 2 times upper limit of normal.
* Administrated of PPI, antibiotic medication within 4 weeks prior to commencement of the study.
* Pregnant and/or lactating women.
* Reproductive aged women not using contraception.
* Uncontrolled diabetics.
* Uncontrolled hypertension.
* Uncontrolled liver dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori as assessed by UBT test | up to 2 months